CLINICAL TRIAL: NCT06796569
Title: Association of Systemic Immune Inflammatory Index with Disease Activity and Lupus Nephritis in Patients with Systemic Lupus Erythematosus
Brief Title: Systemic Immune Inflammatory Index in Systemic Lupus Erythematosus
Status: Recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Shorouk Ayman Mohamed, assistant lecturer, Sohag University
Other Study IDs: soh-Med-25-1-2MD
Record Dates: First submitted 2025-01-22; First posted 2025-01-28 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Systemic Lupus Erythematosus; Lupus Nephritis
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Lupus Nephritis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- patients diagnosed with systemic lupus and lupus nephritis: this group will include 30 patients, all patients will undergo the following: For the evaluation of SLE clinical disease activity SLEDAI ( systemic upus erythematosus disease activity index)scores will be recorded The SII (systemic immune inflammatory index) will be calculatedusing the following formula: SII = (neutrophil count × platelet count)/lymphocyte count.
  Interventions: Diagnostic Test: systemic immune inflammatory index
- patients diagnosed with systemic lupus without lupus nephritis: this group will also include 30 patients, all patients will undergo the following: For the evaluation of SLE clinical disease activity SLEDAI ( systemic upus erythematosus disease activity index)scores will be recorded The SII (systemic immune inflammatory index) will be calculated using the following formula: SII = (neutrophil count × platelet count)/lymphocyte count.
  Interventions: Diagnostic Test: systemic immune inflammatory index
- healthy control group: this group will also include 30 healthy controls , they will undergo the following: The SII (systemic immune inflammatory index) will be calculated using the following formula: SII = (neutrophil count × platelet count)/lymphocyte count.
  Interventions: Diagnostic Test: systemic immune inflammatory index

INTERVENTIONS:
Diagnostic Test: systemic immune inflammatory index — Systemic immune inflammatory index (SII) is a combination of three hematological parameters (platelets, neutrophils, and lymphocytes) and it is calculated using the following formula: SII = (neutrophil count × platelet count)/lymphocyte count.

SUMMARY:
This study aims to investigate the association between the systemic immune-inflammation index and disease activity, as well as lupus nephritis in patients with systemic lupus erythematosus

ELIGIBILITY:
Inclusion Criteria:

* o Older than 16 years

  * In a patient with SLE, patients who fulfill the criteria of the American College of Rheumatology (ACR) and European League Against Rheumatism (EULAR).
  * In patients with LN, patients whose diagnosis is confirmed by kidney biopsy and pathohistological verification (WHO classification, and the International Society of Nephrology/Renal Pathology Society (ISN/RPS) classification.

Exclusion Criteria:

* Patients with other autoimmune rheumatological diseases, lymphoproliferative disorders, malignancies, liver diseases, end-stage kidney disease, diabetic nephropathy, active infections, recent history of blood transfusion and patients with deficiencies in vitamin B12, folate, and iron are excluded from the study.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: patients attending in rheumatology outpatient clinic, sohag university hospital
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2024-12-02 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
association of systemic immune-inflammation index (SII) disease activity in systemic lupus erythematosus | baseline
  This study aims to investigate if there is an association between the systemic immune-inflammation index (SII) and disease activity in patients with systemic lupus erythematosus using SLEDAI(systemic lupus erythematosus disease activity index) as a valid index to compare results with
association of systemic immune-inflammation index (SII) and lupus nephritis in patients with systemic lupus erythematosus | baseline
  This study aims to investigate the association between the systemic immune-inflammation index (SII) and lupus nephritis in patients with systemic lupus erythematosus

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag Faculty, Sohag, Sohag Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No